CLINICAL TRIAL: NCT04359446
Title: Laser-excimer Versus High-pressure Dilation to Treat Under-expansion of the Stent (LASER EXPAND Study)
Brief Title: Laser-excimer Versus High-pressure Dilation to Treat Under-expansion of the Stent
Acronym: LASER EXPAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPIC16- LASER EXPAND
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Diseases; Arterial Disease
Keywords: LASER EXPAND
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Lasers, Excimer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stent under-expansion with NC Balloon (Other)
  Interventions: Procedure: NC ( Non- Compliant) Balloon dilatation
- Stent under-expansion with Laser Excimer + NC Balloon (Other)
  Interventions: Procedure: Laser Excimer + NC Balloon

INTERVENTIONS:
Procedure: NC ( Non- Compliant) Balloon dilatation — NC Balloon dilatation at pressure > NC-RBP (18-20 atm) with > 1 long inflation (> 20 minutes each)
  Arms: Stent under-expansion with NC Balloon
Procedure: Laser Excimer + NC Balloon — Laser Excimer + NC Balloon dilatation at pressure > NC-RBP (18-20 atm) with > 1 long inflation (> 20 minutes each)
  Arms: Stent under-expansion with Laser Excimer + NC Balloon

SUMMARY:
The laser-excimer technology could be an essential tool to correct the under-expansion of the stent once it has been implanted unless severe calcification. The laser-excimer technology achieves a greater minimum luminal area when treating an infra-expanded stent, when compared with the results obtained with the simple dilatation at high or very high pressure.

DETAILED DESCRIPTION:
The laser-excimer technology could be an essential tool to correct the under-expansion of the stent once it has been implanted unless severe calcification.

The investigators propose a study that serves as proof of concept for this technology (laser Excimer) used according to its intended use in this specific substrate of coronary lesions. (stent under-expansion without severe underlying calcification).The laser-excimer technology achieves a greater minimum luminal area when treating an infra-expanded stent, when compared with the results obtained with the simple dilatation at high or very high pressure.

ELIGIBILITY:
Inclusion Criteria:

Patients with:

* Age ≥ 18 years.
* Consecutive real-world patients, referred for cardiac catheterization for any cause, who present in any main vessel, bypass or in the common trunk an under-expanded stent tributary of being treated (minimum luminal area <4 mm2 or <6 mm2 in the left main coronary artery measured by IVUs (Intravascular Ultrasound) / OCT(Optical Coherence Tomography)) and that it is not possible to dilate with a NC balloon to a maximum of 20 atm.

Exclusion Criteria:

* Refusal of the patient to participate in the study.
* Patients with life expectancy <1 year.
* Patients with advanced kidney disease (grade IV) or liver failure (Child C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-09-12 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Variation of the minimum luminal area (MLA) | During procedure
  Detection of rate for Variation of the minimum luminal area (MLA) of the under-expanded stent defined as: ((MLAfinal-MLAinicial) / MLAinicial) x 100.

SECONDARY OUTCOMES:
Hyperacute thrombosis (THA) | During procedure
  Detection of rate for Hyperacute thrombosis defined as: (number of THA patients cases detected / number of total patients cases) x 100.
No- Reflow/Slow Flow (SFL) | During procedure
  Detection of rate for no-reflow / slow flow rate (SFL), defined as (number of detected patients cases of SFL / number total cases) x 100.
Bradycardia | During procedure
  Detection of rate for Bradycardia (HR <50 beats / min or reduction of HR during application> 30%) defined as: (number of detected patients cases of bradycardia / number of total patients cases) x 100.
Tachycardia | During procedure
  Detection of rate for tachycardia, defined as: (ventricular or supraventricular tachycardias detected) during modification of the lesion, defined as (number of patients cases detected / number of total patients cases) x 100.
Procedure time | During procedure
  Determination of the duration time of the procedure in minutes
Contrast Volume | During procedure
  Determination of total contrast volume in mL
Complications during procedure | During procedure
  Detection of rate for complications, defined as: (number of patients cases of coronary perforation, occlusive dissection of the vessel, intra-procedure death, myocardial infarction / total number of cases) x 100.
Periprocedural Infarction complications | During procedure
  Detection of rate for periprocedural infarction complications, defined as: (number of patients cases of periprocedural infarction / total number of patients cases) x 100.

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela, Coruña
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital Universitario Lucus Agusti, Lugo
  - Hospital Universitario La Paz, Madrid

REFERENCES:
- [Background] Byrne RA, Joner M, Kastrati A. Stent thrombosis and restenosis: what have we learned and where are we going? The Andreas Gruntzig Lecture ESC 2014. Eur Heart J. 2015 Dec 14;36(47):3320-31. doi: 10.1093/eurheartj/ehv511. Epub 2015 Sep 28. PMID 26417060
- [Background] Veerasamy M, Gamal AS, Jabbar A, Ahmed JM, Egred M. Excimer Laser With and Without Contrast for the Management of Under-Expanded Stents. J Invasive Cardiol. 2017 Nov;29(11):364-369. PMID 29086727
- [Background] Egred M. A novel approach for under-expanded stent: excimer laser in contrast medium. J Invasive Cardiol. 2012 Aug;24(8):E161-3. PMID 22865316
- [Background] Lam SC, Bertog S, Sievert H. Excimer laser in management of underexpansion of a newly deployed coronary stent. Catheter Cardiovasc Interv. 2014 Jan 1;83(1):E64-8. doi: 10.1002/ccd.25030. Epub 2013 Jul 1. PMID 23703809
- [Background] Egred M, Brilakis ES. Excimer Laser Coronary Angioplasty (ELCA): Fundamentals, Mechanism of Action, and Clinical Applications. J Invasive Cardiol. 2020 Feb;32(2):E27-E35. doi: 10.25270/jic/19.00325. PMID 32005787
- [Background] Latib A, Takagi K, Chizzola G, Tobis J, Ambrosini V, Niccoli G, Sardella G, DiSalvo ME, Armigliato P, Valgimigli M, Tarsia G, Gabrielli G, Lazar L, Maffeo D, Colombo A. Excimer Laser LEsion modification to expand non-dilatable stents: the ELLEMENT registry. Cardiovasc Revasc Med. 2014 Jan;15(1):8-12. doi: 10.1016/j.carrev.2013.10.005. Epub 2013 Oct 22. PMID 24290659
- [Background] Ben-Dor I, Maluenda G, Pichard AD, Satler LF, Gallino R, Lindsay J, Waksman R. The use of excimer laser for complex coronary artery lesions. Cardiovasc Revasc Med. 2011 Jan-Feb;12(1):69.e1-8. doi: 10.1016/j.carrev.2010.06.008. Epub 2010 Oct 20. PMID 21241980